CLINICAL TRIAL: NCT02952300
Title: Comparative Evaluation of Postoperative Pain After Root Canal Preparation With Wave One and Neolix in Acute Irreversible Pulpitis of Mandibular Premolar Teeth
Brief Title: Post Operative Pain of Root Canal Preparation With Wave One and Neolix in Acute Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin hassan youseif, resident at endodontic department faculty of oral and dental medicine CU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-10-146
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Pulpitis - Irreversible
Keywords: irreversible pulpitis; reciprocation; rotation; single file; wave one; neolix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- neolix (Experimental): single full rotation file (Neolix ® Neolix ,France) the first file used is C1 file size 25 taper 12% as orifice opener and for coronal flaring for 2/3 of canal length the A1 file size 25 taper 8% in narrow or curved canals if size 10 K file (Mani Inc., Japan). is passively fit in the canal (most of the canals) , but in case of K-file (Mani Inc., Japan) size 20 loose in the canal so we choose large file size 40 taper 4% either of them to the full working length of the canal
  Interventions: Procedure: neolix
- wave one (Active Comparator): single reciprocating file (Wave One ® Dentsply , Switzerland) the canal preparation is done by primary file size 25 taper 8% in narrow or curved canals if size 10 K file (Mani Inc., Japan) is passively fit in the canal ( most of canals ) , but in case of K-file (Mani Inc., Japan) size 20 loose in the canal so we choose large large file size 40 taper 8% either of them to the full working length of the canal
  Interventions: Procedure: wave one

INTERVENTIONS:
Procedure: neolix — single rotation file
  Arms: neolix
Procedure: wave one — single reciprocation file
  Arms: wave one

SUMMARY:
the aim in this prospective in vivo randomized clinical trial to evaluate the influence of instrumentation technique ( reciprocation single file (wave one ) versus rotation single file (neolix) ) on post operative pain ( incidence ,degree and duration ) after endodontic treatment in single rooted lower premolars with symptomatic irreversible pulpits.

According to the inclusion criteria the patients enrolled in the study and allocated randomly into two groups either Wave One (group A) or Neolix ( group B) the endodontic treatment is done at single visit. firstly the patient's medical and dental history is taken .the patient assign on informed consent. and then,anaesthetized and access cavity performed and root canal preparation is done by either two systems and then irrigation and obturation is done. the patient record the post operative pain in sheet with NRS after 6,12,24,48hr and the operator will recall the patient to check the records and follow up the patient.

DETAILED DESCRIPTION:
Medical and dental history: diagnostic charts will be collected in a case report form by the investigators and confirmed for eligibility with the assistant supervisor.

Radiographic examination : preoperative radiographs will be taken to examine the tooth structure,caries detection , periapical status .

Clinical examination : intraoral examination include visual examination for caries , restoration ,swelling ,fistula . mobility, percussion were done .

Diagnostic criteria for symptomatic irreversible pulpitis:

1. The patient marks moderate to severe pain on the numerical rating scale (NRS) . a horizontal line of 11 marks and 10 intervals each takes numbers from 0 to 10 where 0 = no pain , 1-3 =mild pain , 4-6 = moderate pain , 7-10 = severe pain (recording the baseline degree of pain preoperatively before initiating the endodontic treatment ) all the steps done by the same operator.
2. The patient shows severe pain which lasts long after thermal testing which is done by applying hot compound stick on the tooth after coating it with a lubricant.
3. The patient responds to electric pulp tester at a lower level than the contralateral tooth or the adjacent tooth if the contralateral one is missing.

Intervention:

Forty four patients will included and they will be randomly divided into two groups A =root canal preparation with single reciprocating file (Wave One ® Dentsply , Switzerland) and B = Root canal preparation with single full rotation file (Neolix ® Neolix ,France) each group consisted from 22 patient .

Procedure steps :

1. Patients are asked to rate their pain level on numerical rating scale before the anesthesia injection and the start of the preparation to get the baseline record for the pain preoperatively .
2. The patient will receive inferior alveolar nerve block injections ( 1.8 ml mepivacaine hydrochloride 2% ( 1: 100,000 epinephrine ) using a side loading aspirating syringe and 27-gauge long needle.
3. At 15-minutes post injection, access cavity is performed using round bur size 4 and endo-z bur.
4. Tooth is then isolated using rubber dam to prevent introduction of saliva and Bactria from the oral cavity .
5. Checking the patency of the canal with K- file (Mani Inc., Japan). size 10 taper 0.02, extirpation of pulp with H-file (Mani Inc., Japan). size 15 taper 0.02 .
6. An electronic apex locator ( Morita Corporation, Kyoto, Japan) will be used to determine working length, and then working length will be confirmed radiographically to be adjusted 1mm shorter that the root apex.
7. Each patient has equal chance to enter either the intervention groups A or B group as each patient takes number in excel sheet divided into two groups A and B chosen by assistant supervisor who determine which system will be used with this patient .
8. Comparator group: If the system to by used is Wave One the canal preparation is done by primary file size 25 taper 8% in narrow or curved canals if size 10 K file (Mani Inc., Japan) is passively fit in the canal ( most of canals ) , but in case of K-file (Mani Inc., Japan) size 20 loose in the canal so we choose large large file size 40 taper 8% either of them to the full working length with pre programmed motor (X-Smart Plus (Dentsply) with reducing hand piece 6:1 more anticlockwise angle than clock wise one .
9. Experimental group : If the Neolix systems will be used ,then the first file used is C1 file size 25 taper 12% as orifice opener and for coronal flaring for 2/3 of canal length the A1 file size 25 taper 8% in narrow or curved canals if size 10 K file (Mani Inc., Japan). is passively fit in the canal (most of the canals) , but in case of K-file (Mani Inc., Japan) size 20 loose in the canal so we choose large file size 40 taper 4% either of them to the full working length to the full working length with X-Smart Plus motor with speed 300-500 rpm and torque 1.5 N.cm.
10. Irrigation is made between each file using 2.5% sodium hypochlorite and MD-ChelCream19% ethylenediaminetetraacetic acid cream (METABIOMED company , Korea).
11. The canals are then dried with paper points and obturated with gutta percha and ADSEAL resin sealer(METABIOMED company, Korea) by selection of a master cone corresponding to the size of master apical file, then spreader will be selected to provide auxiliary cones using cold lateral compaction technique.
12. Access cavity is then sealed with temporary filling.
13. then rating of post operative pain after the treatment is recorded by numerical rating scale ( NRS) in sheet given to the patient to record the degree of pain after 6 hrs ,12 hrs ,24 hrs ,48 hrs together with recalling the patient to check the record then the patient return the sheet to the operator and then the collected sheets presented to assistant supervisor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good health(American Society of Anesthesiologists Class II or higher).
2. Patients having symptomatic irreversible pulpitis in one of their mandibular premolars.
3. Age range is between 20 and 35 years.
4. Patients who can understand numerical rating scale (NRS).
5. Patients able to sign informed consent.

Exclusion Criteria:

1. Patients with positive percussion test .
2. Patients having history of necrosis with or without apical pathosis .
3. Patients have sinus tract or fistula extraoral or intraoral.
4. Patients having active pain in more than one pre molar.
5. Patients who had taken analgesics in the 12 hours preceding the preparation.
6. Pregnant or mentally retarded patients.
7. Teeth with grade 2 or 3 mobility.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | up to 48 hours after completion of treatment
  intensity of postoperative pain after treatment by Numerical Rating Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: abeer marouzk, professor, Study Chair — faculty of oral and dental medicine -cairo university; alaa el baz, ass. professor, Study Director — faculty of oral and dental medicine -cairo university; yasmin hassan yousief, resident, Principal Investigator — faculty of oral and dental medicine -cairo university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J. 2008 Feb;41(2):91-9. doi: 10.1111/j.1365-2591.2007.01316.x. Epub 2007 Oct 23. PMID 17956561
- [Background] Tanalp J, Kaptan F, Sert S, Kayahan B, Bayirl G. Quantitative evaluation of the amount of apically extruded debris using 3 different rotary instrumentation systems. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Feb;101(2):250-7. doi: 10.1016/j.tripleo.2005.03.002. Epub 2005 Oct 14. PMID 16448929
- [Background] Nekoofar MH, Sadeghipanah M, Dehpour AR. Evaluation of meloxicam (A cox-2 inhibitor) for management of postoperative endodontic pain: a double-blind placebo-controlled study. J Endod. 2003 Oct;29(10):634-7. doi: 10.1097/00004770-200310000-00005. PMID 14606784
- [Background] Pochapski MT, Santos FA, de Andrade ED, Sydney GB. Effect of pretreatment dexamethasone on postendodontic pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Nov;108(5):790-5. doi: 10.1016/j.tripleo.2009.05.014. Epub 2009 Sep 12. PMID 19748294
- [Background] Ince B, Ercan E, Dalli M, Dulgergil CT, Zorba YO, Colak H. Incidence of postoperative pain after single- and multi-visit endodontic treatment in teeth with vital and non-vital pulp. Eur J Dent. 2009 Oct;3(4):273-9. PMID 19826598
- [Background] Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011 Apr;37(4):429-38. doi: 10.1016/j.joen.2010.12.016. PMID 21419285